CLINICAL TRIAL: NCT05592431
Title: Effect of Volume Guarantee-High Frequency Oscillatory Ventilation on Cerebral Blood Flow in Preterm Neonates
Brief Title: Effect of Volume Guarantee-High Frequency Oscillatory Ventilation on Cerebral Blood Flow in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Abdullah Moussa Akid, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MD 191/2022
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Infant, Premature, Diseases; Respiratory Tract Diseases; Cerebral Blood Flow
Keywords: High Frequency Oscillatory Ventilation; Volume Guarantee-High Frequency Oscillatory Ventilation; Preterm; Cerebral Blood Flow
MeSH Terms: conditions — Infant, Premature, Diseases; Respiratory Tract Diseases; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Frequency Oscillatory Ventilation with Volume Guarantee (HFOV-VG ) (Experimental): After documenting parental consent, preterm neonates with respiratory insufficiency randomly ventilated on (HFOV-VG ) will be assessed by doppler cerebral blood flow velocity measurements
  Interventions: Device: High Frequency Oscillatory Ventilation with Volume Guarantee (SLE6000;SLE)
- High Frequency Oscillatory Ventilation (HFOV) (Active Comparator): After documenting parental consent, preterm neonates with respiratory insufficiency randomly ventilated on (HFOV) will be assessed by doppler cerebral blood flow velocity measurements
  Interventions: Device: High Frequency Oscillatory Ventilation (SLE6000;SLE)

INTERVENTIONS:
Device: High Frequency Oscillatory Ventilation with Volume Guarantee (SLE6000;SLE) — ventilator settings will be recorded such as: inspiratory: expiratory ratio (I:E), fractionated inspired oxygen (FiO2), mean airway pressure (MAP), frequency (HZ), delta P and high-frequency tidal volume (VThf).
  Other Names: transcranial Doppler ultrasonographic examination
  Arms: High Frequency Oscillatory Ventilation with Volume Guarantee (HFOV-VG )
Device: High Frequency Oscillatory Ventilation (SLE6000;SLE) — ventilator settings will be recorded such as: inspiratory: expiratory ratio (I:E), fractionated inspired oxygen (FiO2), mean airway pressure (MAP), frequency (HZ), delta P
  Other Names: transcranial Doppler ultrasonographic examination
  Arms: High Frequency Oscillatory Ventilation (HFOV)

SUMMARY:
A randomized controlled clinical trial evaluates cerebral blood flow changes associated with HFOV-VG in comparison to HFOV alone in preterm neonates with respiratory insufficiency during the period of invasive respiratory support

DETAILED DESCRIPTION:
Neonatal respiratory distress (NRD) is one of the most common problems in the first few days of neonatal life. NRD has been reported to be prevalent in 5 - 29% of the NICU hospitalized neonates.

High-frequency oscillatory ventilation (HFOV) has been used for more than three decades, it is a rescue maneuver for failed conventional mechanical ventilation. It delivers small tidal volumes to improve gas exchange. As it uses a low tidal volume, under the anatomical dead space at supra-physiological respiratory frequencies HFOV can reduce the risk of lung injury related to the ventilator and consequently reduce the risk of bronchopulmonary dysplasia HFOV is indicated for patients with neonatal air leak syndrome, persistent pulmonary hypertension, and meconium aspiration Several factors are known to influence cerebral perfusion during HFOV. Hypercapnia increases cerebral blood flow (CBF) while a reduction in PaCO2 leads to cerebral vasoconstriction and decreases CBF, Hypoxia is also known to increase CBF via cerebral vasodilation HFOV with volume guarantee (HFOV-VG) is a promising new ventilator mode for the treatment of respiratory failure in newborns. HFOV-VG is expected to result in less lung injury since it reduces fluctuations of high frequency tidal volume (VThf), reduces the number of out-of-target pCO2 values and provides fewer hypoxia attacks compared with HFOV alone

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates with gestational age ≤ 35 weeks.
2. Neonates with various causes of respiratory failure: respiratory distress syndrome (RDS), air leak syndromes, pneumonia, or pulmonary hemorrhage, failing with conventional ventilation (i.e. when conventional ventilation failed to maintain either oxygenation or ventilation) and are switched to HFOV as a rescue therapy.

Exclusion Criteria:

1. Preterm neonates with major upper or lower airway anomalies.
2. Preterm neonates with significant congenital anomalies including cardiac, abdominal or respiratory

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Doppler cerebral blood flow velocity measurements | 72 hours
  Investigate the effect of combining the VG mode with HFOV (HFOV-VG), versus the effect of HFOV alone, on Doppler cerebral blood flow velocity measurements

SECONDARY OUTCOMES:
efficiency of HFOV-VG in comparison with HFOV alone | 8 weeks or till patient discharged
  Evaluate the efficiency of HFOV-VG in comparison with HFOV alone as a rescue therapy in providing adequate neonatal ventilation and its possible impact on the short-term clinical outcome in terms of mortality and morbidities of these preterm neonates.
Duration of admission | 8 weeks or till patient discharged
  To document total number of days of admission
Mortality rate | 8 weeks or till patient death which comes first
  To document incidence of mortality during hospitalization
Incidence of feeding intolerance | 8 weeks or till patient discharged
  Percentage of Patients who developed feeding intolerance
Days to reach full intake | 8 weeks or till patient discharge which comes first
  Number of days needed by each patient to reach full intake
Chest x ray change | Before intubation and and after 2 hours on assigned mode
  Chest x ray grading of RDS performed to patient before and after the assigned mode to compare lung aeration degree

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Units (NICUs), Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No